CLINICAL TRIAL: NCT02954809
Title: Feasibility of Bright Light Therapy on Fatigue, Sleep and Circadian Activity Rhythms in Lung Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Oncology Nursing Society (Other)
Responsible Party: Principal Investigator, Carleara Weiss, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 030-702786
Record Dates: First submitted 2016-10-26; First posted 2016-11-03 (Estimated); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Fatigue; Sleep Disturbance; Circadian Dysregulation
Keywords: fatigue; sleep disturbances; circadian activity rhythms
MeSH Terms: conditions — Fatigue; Parasomnias; Chronobiology Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental): Exposure to morning bright light therapy delivered with Green-Blue Re-Timer glasses for 30 minutes in the morning during one week.
  Interventions: Device: Morning bright light therapy
- Attention Control (Active Comparator): Exposure to dim light delivered with Red-Yellow Re-Timer glasses for 30 minutes in the morning during one week.
  Interventions: Device: Dim light

INTERVENTIONS:
Device: Morning bright light therapy — Exposure to morning bright light therapy delivered with Green-Blue Re-Timer glasses for 30 minutes in the morning during one week.
  Arms: Experimental
Device: Dim light — Exposure to dim light with Red-Yellow Re-Timer glasses for 30 minutes in the morning during one week.
  Arms: Attention Control

SUMMARY:
The purpose of this study is to determine the feasibility of a morning bright light therapy intervention for fatigue, sleep disturbances, and circadian activity rhythms in lung cancer survivors.

DETAILED DESCRIPTION:
A randomized controlled trial to test the effects of morning bright light therapy on fatigue, sleep disturbances, and circadian activity rhythms in lung cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III Non-small cell lung cancer survivors
* Must be at >6-weeks and < 3 years post-surgical resection
* Must have diagnosis fatigue and/or sleep disturbances

Exclusion Criteria:

* Individuals clinically unstable.
* Mania, Bipolar disease or seizure disorder
* Macular degeneration or glaucoma.
* Currently receiving chemotherapy or radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dean GE, Redeker NS, Wang YJ, Rogers AE, Dickerson SS, Steinbrenner LM, Gooneratne NS. Sleep, mood, and quality of life in patients receiving treatment for lung cancer. Oncol Nurs Forum. 2013 Sep;40(5):441-51. doi: 10.1188/13.ONF.441-451. PMID 23989018
- [Background] Ancoli-Israel S, Rissling M, Neikrug A, Trofimenko V, Natarajan L, Parker BA, Lawton S, Desan P, Liu L. Light treatment prevents fatigue in women undergoing chemotherapy for breast cancer. Support Care Cancer. 2012 Jun;20(6):1211-9. doi: 10.1007/s00520-011-1203-z. Epub 2011 Jun 11. PMID 21660669
- [Background] Jeste N, Liu L, Rissling M, Trofimenko V, Natarajan L, Parker BA, Ancoli-Israel S. Prevention of quality-of-life deterioration with light therapy is associated with changes in fatigue in women with breast cancer undergoing chemotherapy. Qual Life Res. 2013 Aug;22(6):1239-44. doi: 10.1007/s11136-012-0243-2. Epub 2012 Aug 3. PMID 22865153
- [Background] Ancoli-Israel S, Liu L, Rissling M, Natarajan L, Neikrug AB, Palmer BW, Mills PJ, Parker BA, Sadler GR, Maglione J. Sleep, fatigue, depression, and circadian activity rhythms in women with breast cancer before and after treatment: a 1-year longitudinal study. Support Care Cancer. 2014 Sep;22(9):2535-45. doi: 10.1007/s00520-014-2204-5. Epub 2014 Apr 15. PMID 24733634
- [Background] Redd WH, Valdimarsdottir H, Wu LM, Winkel G, Byrne EE, Beltre MA, Liebman ES, Erazo T, Hayes JA, Isola L, Scigliano E, Meschian Y, Lutgendorf S, Ancoli-Israel S. Systematic light exposure in the treatment of cancer-related fatigue: a preliminary study. Psychooncology. 2014 Dec;23(12):1431-4. doi: 10.1002/pon.3553. Epub 2014 May 2. No abstract available. PMID 24798589

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Attention Control
Started | 7 | 7
Completed | 7 | 5
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Attention Control | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: Total participants that completed study n=12 We recruited 14 participants. Two participants from the attention control group were excluded based on the study exclusion criteria (1) rotating shift work (2) decline in overall health condition/cancer treatment.
  The intent is to report the number of participants who completed the study out of the total enrolled.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 2 | 2 | 4
    >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total participants recruited n=14 Participants that completed study n=12
  Participants
    Female | 5 | 4 | 9
    Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total participants recruited n=14 Participants that completed study n=12
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 7 | 5 | 12
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total participants recruited n=14 Participants that completed study n=12
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 7 | 5 | 12
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Study Completion
Description: The percentage of participants recruited that completed the study
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Attention Control
Number analyzed (Participants) | 7 | 7
Participants | 7 | 5

2. Other Pre Specified Outcome: Changes in Quality of Life With theFunctional Assessment of Cancer Therapy - Lung
Description: Quality of Life will be assessed before, during, and after the intervention.
Time Frame: 5 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Assessment of Environmental Light With Actigraphy (Actiwatch Spectrum Respironics)
Description: Exposure to environmental light will be assessed at pre-test, intervention and post-test for a descriptive analysis
Time Frame: 5 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Assessement of Chronotype With the Morningness Versus Eveningness Questionnaire
Description: Chronotype will be assessed at baseline for a descriptive analysis.
Time Frame: 1 day
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Fatigue Symptoms With Fatigue Severity Index From Pre-test to Post-test
Description: Comparison of fatigue severity from pre-test to post-test.
Time Frame: 5 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Sleep Quality With the Pittsburgh Sleep Quality Index From Pre-test to Post-test
Description: Comparison of Sleep Quality from pre-test to post-test.
Time Frame: 5 Weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes in Insomnia With Insomnia Severity Index From Pre-test to Post-test
Description: Comparison of insomnia from pre-test to post-test.
Time Frame: 5 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Circadian Activity Rhythms With Actigraphy From Pre-test to Post-test
Description: Circadian Activity Rhythms will be assessed with actigraphy during the 5-week time frame.
Time Frame: 5 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Assessment of Visual Acuity With the Snellen Visual Acuity Chart
Description: Visual acuity data will be collected and save for safety purposes only at pre-test and post-test.
Time Frame: 5 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Assessment of Daytime Sleepiness With the Epworth Sleepiness Scale
Description: Daytime Sleepiness will be assessed for safety purposes only at pre-test, intervention and post-test. Individuals with high daytime sleepiness and/or at risk of falling asleep while driving or performing hazardous activities will be referred out to primary care
Time Frame: 5 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Although no adverse events were reported in this study, anticipated adverse events included eye strain and headache.
Arm/Group | Experimental | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT02954809/Prot_SAP_000.pdf